CLINICAL TRIAL: NCT02333357
Title: Multimedia Toolkits to Implement 12-Step Recovery Concepts in Group Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0905; R01AA017867 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2015-01-07 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Abuse; Drug Abuse
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toolkit (Experimental): Counselors randomized to the toolkit (TK) condition will receive a one to three hour standardized toolkit orientation that will include a description of the overall goal of the toolkit curriculum comprised of five modules, the purpose of each individual element of the toolkit, and an introduction to the toolkit teaching aids such as counselor guides, posters, and patient materials (hand-outs, sampling menus, worksheets, etc). TK counselor participants then conduct group treatment sessions using the toolkit materials with their patient participants.
  Interventions: Behavioral: Multimedia 12-Step Toolkit
- Treatment as Usual (Active Comparator): Counselors assigned to the Treatment as Usual (TAU) attention control condition complete a training that reviews the same five 12-step topics that are included in the toolkit, but they do not receive any toolkit materials. TAU counselor participants then conduct group treatment sessions on the 12-step topics without using toolkit materials.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Multimedia 12-Step Toolkit — The Multimedia 12-Step Toolkit includes counselor written guides, posters, client worksheets, engagement activities, and videos designed to be shown during group treatment sessions to explain and encourage 12-step participation.
  Arms: Toolkit
Behavioral: Treatment as Usual — Treatment as Usual is defined as five standard 12-step facilitation group sessions as counselors would normally conduct with their clients.
  Arms: Treatment as Usual

SUMMARY:
This study is developing and testing a 12-step toolkit with five modules, training counselors to use them, and studying their frequency of use, desirability, effectiveness and patient outcomes. The toolkit includes counselor written guides, posters, client worksheets, engagement activities, and videos designed to be shown during substance abuse treatment group sessions to explain and encourage 12-step participation.

DETAILED DESCRIPTION:
The study has three aims. Aim 1 involves the development of an evidence-based 12-step facilitation toolkit curriculum. Toolkit structure and content is grounded in theory and empirical findings, and incorporates feedback from 12-step facilitation experts and individuals with a history of substance abuse. Aim 2 consists of implementing the resulting five-module Toolkit in a multi-site randomized controlled trial using a pre-/post-Toolkit training design that includes 1- and 6-month post-training assessments. Group counselors employed at community-based outpatient and inpatient substance abuse treatment programs will be randomly assigned to a Toolkit or treatment-as-usual condition. Data obtained from audiotaped sessions will identify between group differences in counselor adherence to 12-step content and skillfulness. Additional data will be collected on counselor satisfaction, 12-step attitudes and beliefs, and 12-step knowledge, as well as on Toolkit acceptability, feasibility, and short-term sustainability. Aim 3 will determine whether exposure to the Toolkit curriculum results in stable 12-step involvement and decreased self-reported substance use among clients.

ELIGIBILITY:
Inclusion Criteria for Counselors:

* Over 18 years of age
* Employed at a participating substance abuse treatment facility
* Provide treatment in a group format

Exclusion Criteria for Counselors:

* At the time of the project they do not have primary responsibility for conducting at least three substance abuse group sessions per week
* Their therapy group is normally scheduled to run less than 50 minutes, or more than 150 minutes
* Unable to provide valid informed consent

Inclusion Criteria for Clients:

* Over 18 years of age
* Attending an observed group of a participating counselor
* (For participation in the Follow-Up Study/Aim 3 only) patients must endorse heavy drinking, alcohol-related difficulties, or poor prior 12-step participation

Exclusion Criteria for Clients:

- Unable to provide valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3483 (Actual)
Dates: Start 2011-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in counselor content adherence from baseline, as measured by the Group Observation Rating System | 0, 1, 6 months
  Counselor adherence to 12-step concepts covered in group sessions assessed using the Group Observation Rating System which consists of items designed to assess general counseling competency skills and 12-step facilitation items
Change in counselor therapeutic skillfulness from baseline, as measured by the Group Observation Rating System | 0, 1, 6 months
  Counselor therapeutic skillfulness when delivering 12-step content in group sessions assessed using the Group Observation Rating System which consists of items designed to assess general counseling competency skills and 12-step facilitation items

SECONDARY OUTCOMES:
Change in counselor satisfaction from baseline, as measured by the Counselor Satisfaction Form | 0, 1, 6 months
  Counselor satisfaction with their group sessions as measured by the Counselor Satisfaction Form which assesses counselors' overall satisfaction with the five 12-step groups
Change in counselor 12-step attitudes and beliefs from baseline, as measured by the Counselor 12-Step Attitudes and Beliefs Scale | 0, 1, 6 months
  Counselor attitudes and beliefs about 12-step recovery and self-help approaches as measured by the Counselor 12-step Attitudes and Beliefs Scale (C-TAB) which queries about current 12-step referral practices, attitudes and beliefs about 12-step recovery and self-help approaches in general, strategies used to assist clients in engaging in the 12-step fellowship, and level of agreement with specific statements about 12-step groups
Change in counselor 12-step knowledge from baseline, as measured by the Counselor Core Elements of 12-step Knowledge Inventory | 0, 1, 6 months
  Counselor knowledge about 12-step concepts as measured by the Counselor Core Elements of 12-step Knowledge Inventory (C-CETSKI), which focuses on the five toolkit content areas
Change in counselor feasibility and sustainability of the toolkit from baseline, as measured by a bi-weekly web-based calendar | 0, 1, 6 months
  Feasibility and short-term sustainability will be measured via a web-based calendar which measures the type and frequency of the 12-step topics and toolkit materials counselors have used
Change in client involvement in 12-step activities from baseline, as measured by the Patient AA Attendance and Involvement Scale | 0, 2, 4, 12, 24 weeks
  Number of 12-step meetings attended and engagement in other 12-step activities as measured by the Patient AA Attendance and Involvement Scale (PAIS) which assesses 12-step recovery activities
Change in client substance use from baseline, as measured by the Substance Use Inventory | 0, 2, 4, 12, 24 weeks
  Self-reported alcohol and drug use as measured by the Substance Use Inventory (SUI), which is a modification of the Time-Line Follow-back Method in which a rater elicits frequency (in days) of consumption of alcohol and other illicit drugs as well as an estimate of average intensity of use

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly C Kirby, PhD, Principal Investigator — Treatment Research Institute
Locations (11):
- United States (11):
  - Genesis Counseling Centers, Camden, New Jersey
  - Phoenix House, Brooklyn, New York
  - Eagleville Hospital, Eagleville, Pennsylvania
  - Livengrin Foundation, Levittown, Pennsylvania
  - Rehab After Work, Philadelphia, Pennsylvania
  - Penn Presbyterian, Philadelphia, Pennsylvania
  - Self-Help Movement, Philadelphia, Pennsylvania
  - Sobreity Through Outpatient, Philadelphia, Pennsylvania
  - The Kirkbride Center, Philadelphia, Pennsylvania
  - The Wedge Recovery Centers, Philadelphia, Pennsylvania
  - Gaudenzia Inc., Philadelphia, Pennsylvania